CLINICAL TRIAL: NCT00895297
Title: Phase II Efficacy and Safety Study of Dasatinib in Patients With Chronic and Accelerated Phase Chronic Myeloid Leukemia Relapsing After Allogeneic Blood or Bone Marrow Transplantation
Brief Title: Efficacy and Safety Study of Dasatinib in Patients With Chronic Myeloid Leukemia
Acronym: Dasatinib
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow recruitment. No safety concerns during this study.
Sponsor: European Society for Blood and Marrow Transplantation (Network)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Ruzena Uddin, EBMT
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2008-001361-29; CLWP-001-2008 (Other: EBMT)
Record Dates: First submitted 2009-05-06; First posted 2009-05-08 (Estimated); Last update posted 2011-12-07 (Estimated); Status verified 2011-12

CONDITIONS: Chronic Myeloid Leukemia
Keywords: Relapsing after allogeneic transplantation; Dasatinib; Sprycel; Philadelphia Chromosomes
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — Dasatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Dasatinib (Sprycel) — 100mg of Dasatinib will be administered as tablets, by mouth, once a day (or twice in some cases depending on the stage of the disease) consistently either in the morning or evening for 12 months. Dose of Dasatinib will be modified according to the patients response.

SUMMARY:
This is a phase II efficacy (indicates the capacity for beneficial change or therapeutic effect) and safety study of Dasatinib in patients with relapsed Chronic Myeloid Leukemia (CML) following a Stem Cell Transplant (SCT) and who are not benefiting from other treatment, such as imatinib therapy.

A relapse is when an illness that has seemed to be getting better, or to have been cured, comes back or gets worse again.

A total of 50 patients ≥18 years of age will be registered on the trial.

DETAILED DESCRIPTION:
Primary Objective:

1. To assess the efficacy of Dasatinib therapy in chronic and accelerated phase BCR-ABL (+) (Ph + and Ph -) CML patients that undergo molecular, cytogenetic or haematological relapse following SCT.

Secondary Objective(s):

1. To assess the impact of Dasatinib therapy on patient survival after relapse post-SCT and the incidence of any subsequent need for 'rescue' DLI.
2. To assess the safety of Dasatinib in this clinical context using this specific dose regimen

Chronic myeloid leukaemia (CML) is a form of cancer that starts in cells within the bone marrow called haematopoietic stem cells. Stem cells are immature cells which can divide many times and eventually produce all the lymphocytes and myeloid cells present in the blood. They are produced in the bone marrow - the spongy tissue found in large bones, including the pelvis, sternum, limb bones and the ribs.

Leukaemia is a cancer of the white blood cells. In CML, too many myeloid cells (one of the main types of white blood cells which defend the body against infectious diseases) are produced. The myeloid cells are released into the blood when they are immature and unable to work properly. These immature white blood cells are known as blasts.

The immature cells fill up the bone marrow and prevent it from making blood cells properly. As the leukaemia cells do not mature, they can't do the work of normal white blood cells, which leads to an increased risk of infection. Because the bone marrow is overcrowded with immature white cells it also can't make enough healthy red cells and platelets.

CML usually develops very slowly, which is why it is called 'chronic' myeloid leukaemia.

The aim of this study is to assess the efficacy (indicates the capacity for beneficial change or therapeutic effect) of a leukaemia treatment called dasatinib (sprycel) in patients with relapsed Chronic Myeloid Leukaemia (CML) following a Stem Cell Transplant (SCT) and who are not benefiting from other treatment, such as imatinib therapy.

A relapse is when an illness that has seemed to be getting better, or to have been cured, comes back or gets worse again.

Dasatinib works by blocking (inhibiting) signals within cancer cells that cause the cell to grow and divide.

The growth of cells in our bodies is controlled by signals that switch on and off within the cells. When the signals for growth are switched on the cells are triggered to grow and multiply. People with CML have an abnormal signaling protein inside their leukaemia cells. This abnormal protein sends out grow-and-divide signals to the cells at all times and never switches off.

Dasatinib finds the faulty protein and locks onto it. This prevents the protein from stimulating the cells to grow. Dasatinib is known as a signal transduction inhibitor, because it blocks the 'grow' signal. The chemical it blocks is called tyrosine kinase, so dasatinib is also known as a tyrosine kinase inhibitor.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients greater or equal to 18 years of age.
2. Diagnosed with BCR-ABL (+) Chronic Myeloid Leukemia (they can be Philadelphia chromosome positive or negative)
3. Prior therapy including imatinib
4. Patients transplanted from an HLA-identical sibling or an HLA-matched unrelated donor.
5. Patients transplanted in first chronic phase or accelerated phase.
6. Patients with untreated relapse of BCR-ABL (+) CML (they can be Philadelphia chromosome positive or negative) after allogeneic transplantation and entered within 6 weeks of the first detection of relapse.
7. Molecular, cytogenetic or haematological relapse in chronic or accelerated phase.
8. Written informed consent.
9. Absence of serious concomitant illness

Exclusion Criteria:

1. Patients relapsing in blast crisis.
2. Patients transplanted after blastic transformation of CML.
3. Patients receiving any therapy for relapse other than withdrawal of immunosuppression (DLI is not permitted).
4. Patients treated with other investigational agents during the previous 30 days
5. Patients previously treated with Dasatinib.
6. Absence of written informed consent.
7. Presence of serious concomitant disease.
8. History of a significant bleeding disorder unrelated to CML.
9. Pregnancy or lactation status positive.
10. SGOT and SGPT more than 2.5 x the upper limit of the normal range as determined by the laboratory where the analysis is performed.
11. Total serum bilirubin level more than 2 x the upper limit of the normal range of the laboratory where the analysis is performed.
12. Serum creatinine concentration more than 1.5 x the upper limit of the normal range of the laboratory where the analysis is performed.
13. Concomitant Medications, any of the following should be considered for exclusion:

    * Category I drugs that are generally accepted to have a risk of causing Torsades de Points including: (Patients must discontinue drug 7 days prior to starting Dasatinib):
    * quinidine, procainamide, disopyramide.
    * amiodarone, sotalol, ibutilide, dofetilide.
    * erythromycin, clarithromycin.
    * chlorpromazine, haloperidol, mesoridazine, thioridazine, pimozide, ziprasidone.
    * cisapride, bepridil, droperidol, methadone, arsenic, chloroquine, domperidone, halofantrine, levomethadyl, pentamidine, sparfloxacin, lidoflazine.
    * The concomitant use of H2 blockers or proton pump inhibitors with Dasatinib is not recommended. The use of antacids should be considered in place of H2 blockers or proton pump inhibitors in patients receiving Dasatinib therapy. If antacid therapy is needed, the antacid dose should be administered at least 2 hours prior to or 2 hours after the dose of Dasatinib.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2010-02; Primary Completion 2011-10 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
CMR as determined by two consecutive (-) RT-PCR tests for the presence of BCR-ABL transcripts in peripheral blood samples 1 year after starting Dasatinib therapy. The expected CMR of >30% would be regarded as being clinically relevant | 4 years

SECONDARY OUTCOMES:
Complete haematological response (CHR) at 3 months post commencing Dasatinib for those that have relapsed at the haematological level. | 4 years
Complete cytogenetic response (CCyR) at 6 and 12 months post commencing Dasatinib for those that have relapsed at the cytogenetic level. | 4 years
Major molecular response (MMR) at 12 months post commencing Dasatinib for all patients. | 4 years
Proportion of patients requiring DLI during the first 12 months | 4 years
Overall survival (OS) - Limited to 3 years. | 4 years
Progression free survival (PFS). | 4 years
Adverse event (AE) rate. | 4 years
Rate of dose reductions, interruptions and discontinuations. | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo L Olavarria, Dr, Principal Investigator — Hospital De Navarra Irunlarrea, Spain
Locations (7):
- E Herriot Hospital, Lyon, France
- Germany (3):
  - University Hospital, Hamburg
  - Uniklinik Leipzig, Leipzig
  - Stiftung Deutsche Klinik für Diagnostik, Wiesbaden
- Switzerland (2):
  - University Hospital, Basel
  - Hopitaux Universitaires de Geneve, Geneva
- Hammersmith Hospital, London, United Kingdom

REFERENCES:
- See also: Sponsor website — http://www.ebmt.org